CLINICAL TRIAL: NCT04638296
Title: Perceptions On Music And Noise In The Operating Room: A Cross Sectional Study
Brief Title: Perceptions On Music And Noise In The OR
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Rana Sharara, Associate Professor of Clinical Pediatrics and Pediatric Critical Care, American University of Beirut Medical Center
Other Study IDs: SBS-2018-0310
Record Dates: First submitted 2020-11-09; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-11

CONDITIONS: Noise Exposure; Surgical Procedure, Unspecified; Physician's Role; Nurse's Role; Performance Anxiety; Concentration Ability Impaired
Keywords: Music; Operating Room; Noise; Surgery
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians: surgeons, anesthesiologists, and surgical residents
  Interventions: Other: Interviews
- Nurses: OR Nurses
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — The investigators designed 3 versions of the semi structured interview guide for each of the surgeons/anesthesiologists (Appendix A.1), residents (Appendix A.2) and nurses (Appendix A. 3). All versions were subdivided into 3 general categories: 1) participant demographics such as participant's age, years of experience, specialty, years of employment at the institution 2) participant's perceptions of noise in the OR, what they considered as sources of noise, the loudness level, whether they thought this impacted their concentration, performance, communication, whether this was distracting or helpful in different stages of the operation, and 3) perceptions on music.

SUMMARY:
Background: Noise in operating rooms (ORs) during surgery may affect OR personnel and pose a threat to patient safety. The sources of noise vary depending on the operation. We aimed to study how OR staff perceived noise, whether music was considered noise and what its perceived effects were.

Methods: Surgeons, anesthesiologists, residents, and nurses were interviewed. IPads were placed in the ORs to gather noise level data.

DETAILED DESCRIPTION:
1. Introduction

   High noise levels in the operating rooms (ORs) during surgery may pose a major threat to the safety and efficiency of procedures performed [1]. The recommended threshold for noise should not exceed 90 dBA over an 8 hour period to prevent noise induced hearing loss [2]. Unfortunately, in 40% of surgeries, OR noise levels reach and exceed 100-120 dBA [2], comparable to a busy highway (1). High noise levels affect both patients and staff: patients may suffer from intraoperative hypertension and tachycardia [3], and prolonged exposure of staff to OR noise has been linked to noise induced hearing loss [4,5], to interference with communication in the OR (6) and to decrements in surgeons' concentration and vigilance [4,7,8].

   Sources of noise in the OR stem primarily from (a) surgical instruments including high speed pneumatic drills, chisels, hammers, and saws [9], (b) equipment such as vital sign monitors, alarms, ventilators, anesthesia machines, waste management devices, and radiological equipment [6] and (c) conversations amongst the staff [4]. Clanging, clattering or dropping metal instruments is also another source of noise [1]. In addition to the above, music is occasionally played in ORs, often requested and chosen by the operating surgeon; whether music qualifies as just more noise is debatable [5]. There have been mixed reports on the effect of music on personnel performance, concentration, communication, speed and cooperation [8, 10-16]. Proponents of music claim that it masks some of the noise, has a calming effect, improves motivation, increases accuracy, and reduces stress [1, 11, 12, 14, 15, 17]. A review of the literature describes the effect of music as contributing to overall stress of the environment, interfering with communication, and posing a threat to the safety of patient and staff as well as to task completion [5].

   The literature is lacking in research on the effects of music as a distractor during operations, especially given the likelihood of unexpected stressful intraoperative complications [18]. It is not clear if at a critical time in a race against the clock, music incentivizes the surgeon and OR staff or if it exacerbates their stress and distracts them.

   Our aim was to determine how surgeons, anesthesiologists, residents and nurses perceived the presence of noise and music in the operating room and how they thought it affected their performance, concentration and communication. The results of this study will guide the design of a follow up study to determine the effects of music on outcomes of specific procedures.
2. Material and Methods 2.1 Study design and setting:

This was an observational, cross sectional study between January 2019-January 2020 of OR personnel's perceptions of noise and music in the ORs at a tertiary academic institution in Beirut, Lebanon. Interviews were conducted in the privacy of the physician's lounge or in a private location within the hospital at the participant's convenience. IPads were placed in all of the center's ten ORs. They were placed in the corner of the ORs away from the working areas and mounted on the walls to avoid interference with the work of the staff.

This research is reported in line with the STROCSS guideline [19].

2.2 Participants:

All OR staff were eligible for recruitment, including surgeons, anesthesiologists, residents and nurses. There were no exclusion criteria per se; however, the interview had to be conducted on the day the participant was involved in a surgical operation.

2.3 Sample Size:

The sample size was estimated at 85 participants. This value was based on a correlation sample size calculation, with a Type I error rate of 0.05, Type II error rate of 0.2, and an expected correlation coefficient of 0.3. Data for this study was collected from 91 participants to err on the side of caution and to maintain heterogeneity among the different staff groups.

2.4 Recruitment:

Participants were recruited via a scripted invitation email detailing the specifics of the study sent by the IT Academic Core Processes and Systems (ACPS) on behalf of the investigating team per ethical research conduct guidelines. Willing potential participants were asked to contact the study team for any questions and to schedule a private meeting for the interview at their convenience. Participation was entirely voluntary, and interviews were conducted following the participants' explicit written consent. Some interviews were audio recorded following participant's consent; otherwise, the interviewer took notes. Interviews lasted approximately 20 minutes.

2.5 Instruments:

Semi Structured Interview Guide The investigators designed 3 versions of the semi structured interview guide for each of the surgeons/anesthesiologists.1), residents and nurses . 3). All versions were subdivided into 3 general categories: 1) participant demographics such as participant's age, years of experience, specialty, years of employment at the institution 2) participant's perceptions of noise in the OR, what they considered as sources of noise, the loudness level, whether they thought this impacted their concentration, performance, communication, whether this was distracting or helpful in different stages of the operation, and 3) perceptions on music.

Most questions were closed ended: effects of noise/music on concentration, performance and communication, and levels of loudness. Answers were rated on 3- point Likert scales (3-Positively, 2- Neutral, 1-Negatively and 3-High, 2- Moderate, 1- Low, respectively). These were followed by open ended questions referring to the potential effects of noise and music: 1. At which times during surgery do you find music helpful, and why? and 2. At which times during surgery do you find music distracting? Answers to these questions were reviewed and collated thematically.

IPads IPads installed in the ORs were placed in a thin plastic bag in the corner of each operating room. This is to ensure that the iPads did not interfere with the work of the staff. The iPads were iPad Air Wi-Fi 64 GB. The application "Sound Affects" was installed on the iPads and used to extract the noise data. The application was developed by Memac Ogilvy for the institution based on technical requirements from the Patient Affairs Unit. It uses the built in microphone of the iPad hence accounting for the relative loudness perceived by the human ear, which is known as A-weighting value.

2.6 Statistical Analyses:

Quantitative data from interviews was entered into the Statistical Package for Social Sciences (SPSS) version 24 (IBM Corp.) for analysis. Descriptive analyses were carried out using the number and percent for categorical variables and mean and standard deviation for continuous variables and analyzing the noise level data gathered from the sensors and iPads. Pearson Chi square and correlation tests were performed to test for relationships. Narrative responses to open ended questions were categorized thematically.

ELIGIBILITY:
All OR staff were eligible for recruitment

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All OR staff were eligible for recruitment, including surgeons, anesthesiologists, residents and nurses. There were no exclusion criteria per se; however, the interview had to be conducted on the day the participant was involved in a surgical operation.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Perceptions on Noise in the OR | 1 year
  Via an interview participants were asked about their perception on noise in the OR, the sources of noise and how it affected their performance, concentration and communication.
Perceptions on Music in the OR | 1 year
  Via an interview participants were asked about their perception on music in the OR, the sources of noise and how it affected their performance, concentration and communication.

CONTACTS AND LOCATIONS:
Locations (1):
- American University of Beirut Medical Center, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No